CLINICAL TRIAL: NCT01726387
Title: Self-Management Support in Primary Care
Brief Title: Self-Management for Anxiety, Depression and Somatoform Disorders
Acronym: SMADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMADS
Record Dates: First submitted 2012-11-03; First posted 2012-11-14 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Anxiety Depression (Mild or Not Persistent); Major Depressive Disorder, Single Episode, Unspecified; Neurotic, Stress-related and Somatoform Disorders
MeSH Terms: conditions — Lymphoma, Follicular; Depressive Disorder, Major; Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychosocial Counseling (Experimental): A Counseling Assistant offers a low-threshold intervention (self-management support, counseling, active guidance). This nurse practitioner collaborates extensively with the general practitioner, re-adjusting the intervention in order to meet the patient's needs.
  Interventions: Behavioral: Psychosocial Counseling
- Usual Care (Placebo Comparator): Depending on the conditions, patients get usual care of their general practitioner.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Psychosocial Counseling — Depending on their condition, counseling assistants support patients in self-management support, enhancing self-efficacy, reducing psychological symptoms
  Other Names: Minimal Psychological Intervention; Self-Management Support
  Arms: Psychosocial Counseling
Behavioral: Usual Care — Depending on the conditions, patients get usual care of their general practitioner
  Arms: Usual Care

SUMMARY:
Anxiety, Depression and Somatoform disorders are highly prevalent in primary care. Very often these conditions remain undiscovered and/or untreated.

In order to ease this urgent health care problem in the future, the investigators conduct a cluster-randomized controlled trial, implementing a tandem working cooperation between a nurse practitioner (Counseling Assistant - CA) and a general practitioner (GP) on-site its own practise.

The CA's task is to enhance the patients abilities to engage in a better self-management of their psychological symptoms and complaints, to enhance self-efficacy and empower the patients to tackle problems of daily living.

DETAILED DESCRIPTION:
Anxiety, Depression and Somatoform disorders are highly prevalent in primary care. Very often these conditions remain undiscovered and/or untreated. Managing it is time-consuming and communication-intensive. Furthermore, the management is restraint by the high contact-frequencies in primary care practices in Germany.

In order to ease this urgent health care problem in the future, the investigators conduct a cluster-randomized controlled trial, implementing a tandem working cooperation between a nurse practitioner (Counseling Assistant - CA) and a general practitioner (GP) on-site its own practise.

The CA's task is to enhance the patients abilities to engage in a better self-management of their psychological symptoms and complaints, to enhance self-efficacy and empower the patients to tackle problems of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Patients scoring >= 5 on the Patient Health Questionnaire (German Version), corresponding to a probable or established diagnosis of Anxiety, Depression or Somatoform Disorder

Exclusion Criteria:

* Negation of Inclusion Criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
General Self-Efficacy Scale (GSE) | Baseline, 8 Weeks, 12 Months
  GSE assesses a general sense of perceived self-efficacy. It predicts coping with daily hassles as well as adaptation after experiencing all kinds of stressful life events.
  http://userpage.fu-berlin.de/%7Ehealth/engscal.htm "The construct of Perceived Self-Efficacy reflects an optimistic self-belief (Schwarzer, 1992). This is the belief that one can perform a novel or difficult tasks, or cope with adversity -- in various domains of human functioning. Perceived self-efficacy facilitates goal-setting, effort investment, persistence in face of barriers and recovery from setbacks. It can be regarded as a positive resistance resource factor. Ten items are designed to tap this construct. Each item refers to successful coping and implies an internal-stable attribution of success. Perceived self-efficacy is an operative construct, i.e., it is related to subsequent behavior and, therefore, is relevant for clinical practice and behavior change."

SECONDARY OUTCOMES:
Change in Symptom Score Patient's Health Questionnaire (German Version) | Baseline, 8 Weeks, 12 Months
  Reducing the symptoms score in the "Patient's Health Questionnaire (German Version)". Reducing symptom score per scale -2,5 units comparing group mean of the intervention group and the group mean of the control group, power 80%, probability 0,05. Effect size d=0,5.
Health Related Quality of Life | Baseline, 8 Weeks, 12 Months
  Enhancing the health related quality of life in the patients using EQ-5D
  http://www.euroqol.org/ EQ-5D (European-Quality-of-Life-5-Dimensions): "Descriptive system of health-related quality of life states consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of three responses. The responses record three levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension."

OTHER OUTCOMES:
Coping with Illness scale | Baseline, 8 Weeks, 12 Months
  Assesses a broad range of cognitive, behavioral and emotional aspects of coping with illness. Investigators use the short version (FKV-LIS)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Scherer, Prof., Principal Investigator — UK Hamburg-Eppendorf (Germany), Department of Primary Medical Care
Locations (1):
- Primary Care Practices, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zimmermann T, Puschmann E, Ebersbach M, Daubmann A, Steinmann S, Scherer M. Effectiveness of a primary care based complex intervention to promote self-management in patients presenting psychiatric symptoms: study protocol of a cluster-randomized controlled trial. BMC Psychiatry. 2014 Jan 3;14:2. doi: 10.1186/1471-244X-14-2. PMID 24387048
- [Background] Zimmermann T, Puschmann E, Bäter G, Carstens S, Scherer M. Selbstmanagement stärken bei psychosozialen Belastungen. Die Kerbe - Forum für soziale Psychiatrie 4, 24-26, 2012.
- [Background] Zimmermann T, Puschmann E, Porzelt S, Ebersbach M, Ernst A, Thomsen T, Scherer M. Selbstmanagementförderung in der ambulanten Versorgung. Programm einer niedrigschwelligen, komplexen, psychosozialen Intervention durch Pflegekräfte in der Hausarztpraxis. Zeitschrift für Allgemeinmedizin, 91, 11, 456-462, 2015.
- [Background] Porzelt S, Zimmermann T, Ernst A, Puschmann E, Scherer M. Wie Pflegekräfte in der hausärztlichen Versorgung Patienten mit psychischen Beschwerden gezielt unterstützen können. Pflegewissenschaft, 18(7-8): 355-361, 2016.
- [Result] Zimmermann T, Puschmann E, Porzelt S, Ebersbach M, Ernst A, Thomsen P, Scherer M. [Promoting Self-Management in Primary Care - the Association of Motivation for Change, Self-Efficacy and Psychological Distress Prior to the Onset of Intervention]. Psychiatr Prax. 2015 Jul;42 Suppl 1:S44-8. doi: 10.1055/s-0034-1387686. Epub 2015 Jul 2. German. PMID 26135280
- [Result] Zimmermann T, Puschmann E, van den Bussche H, Wiese B, Ernst A, Porzelt S, Daubmann A, Scherer M. Collaborative nurse-led self-management support for primary care patients with anxiety, depressive or somatic symptoms: Cluster-randomised controlled trial (findings of the SMADS study). Int J Nurs Stud. 2016 Nov;63:101-111. doi: 10.1016/j.ijnurstu.2016.08.007. Epub 2016 Aug 21. PMID 27611093
- [Result] Grochtdreis T, Zimmermann T, Puschmann E, Porzelt S, Dams J, Scherer M, Konig HH. Cost-utility of collaborative nurse-led self-management support for primary care patients with anxiety, depressive or somatic symptoms: A cluster-randomized controlled trial (the SMADS trial). Int J Nurs Stud. 2018 Apr;80:67-75. doi: 10.1016/j.ijnurstu.2017.12.010. Epub 2017 Dec 29. PMID 29353712